CLINICAL TRIAL: NCT06075758
Title: Real-World Evidence Study for the Safety and Effectiveness of Ribociclib in Combination With Hormonal Therapy in Patients With HR+/HER2- Advanced or Metastatic Breast Cancer in the Middle East Region
Brief Title: A Study of Ribociclib in Combination With Hormonal Therapy in HR+/HER2- Advanced or Metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AIC01
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: HR+/HER2- advanced/metastatic breast cancer; NIS; Ribociclib; Middle eastern countries
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- ribociclib ambispective: Ambispective patients should have initiated Ribociclib, in combination with hormonal therapy, for at least 12 months before the patient's recruitment date and are still on Ribociclib in combination with hormonal therapy at recruitment. These patients will be followed up till progression, death, Ribociclib discontinuation due to adverse events, or till a maximum period of 6 months, whichever comes first.
  Interventions: Other: ribociclib
- ribociclib retrospective: Retrospective patients should have been on Ribociclib in combination with hormonal therapy for at least 18 months and stopped the medication before the patient's recruitment
  Interventions: Other: ribociclib

INTERVENTIONS:
Other: ribociclib — There is no treatment allocation for NIS trials, patients on administered ribociclib by prescription will be enrolled.
  Treatment plan represents the prescription.
  Other Names: CLEE011

SUMMARY:
This is a non-interventional, ambispective, observational cohort study describing the real-world safety data of approximately 550 Hormone receptor / Human epidermal growth factor receptor 2 (HR+/HER2-) advanced/metastatic breast cancer patients who have received ribociclib combined with hormonal therapy in pre-and postmenopausal women or men in Middle Eastern countries.

DETAILED DESCRIPTION:
The investigators will have a six-month recruitment period to include the eligible subjects as per the protocol selection criteria. Retrospective patients should have been on Ribociclib in combination with hormonal therapy for at least 18 months and stopped the medication before the patient's recruitment.

Ambispective patients should have initiated Ribociclib, in combination with hormonal therapy, for at least 12 months before the patient's recruitment date and are still on Ribociclib in combination with hormonal therapy at recruitment. These patients will be followed up till progression, death, Ribociclib discontinuation due to adverse events, or till a maximum period of 6 months, whichever comes first.

Data will be collected from patient electronic medical records in the sites chosen for patients who received Ribociclib, in combination with hormonal therapy, in the first or second-line setting available in the relevant institutions.

A total of 550 patients is planned for this study. The planned sample size should capture very common adverse events reported in previous studies as well as adverse events ≥ 10% occurring in grade 3 and grade 4 with precision ±2.5%.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years old at the time of receiving Ribociclib in combination with hormonal therapy.
2. Advanced /metastatic breast cancer
3. Estrogen-receptor-positive and/or progesterone receptor-positive breast cancer.
4. HER2-negative breast cancer.
5. Patients who received or currently receiving Ribociclib in combination with hormonal therapy in the first or second-line settings as per the routine practice.
6. For the ambispective part, patients should have initiated the Ribociclib, in combination with hormonal therapy, line of treatment at least 12 months before the patient's recruitment date and still continuingcontinuing the drug at the baseline visit.
7. For retrospective patients only, the patients should have been on Ribocilib, in combination with hormonal therapy, for at least 18 months and stopped Ribociclib before the SIV date.enrollment
8. For ambispective part, patients agree to sign informed consent before their enrollment.

Exclusion Criteria:

1. Ribociclib-based treatment regimen beyond the second line.
2. Patients are currently participating in any other clinical trials.
3. Patient with a known hypersensitivity to any of the excipients of Ribociclib.
4. Patients who previously received any other CDK4/6 inhibitor .
5. For ambispective patients, patients who refuse to sign the informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- advanced/metastatic breast cancer patients who have received Ribociclib in combination with hormonal therapy in pre-and postmenopausal women or men in Middle Eastern countries
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
AEs/SAEs/ severity and frequency | 18 months
  Frequency/ severity of adverse events and lab abnormalities of HR+/HER2- advanced/metastatic breast cancer patients who have received Ribociclib in combination with hormonal therapy at 6and 18 months.

SECONDARY OUTCOMES:
Proportion of patients who are progression-free | 6 months, 18 months
  Percentage of progression-free patients (at 18 months following the start date of ribociclib and at the end of ribociclib treatment),
Proportion of patients with clinical benefit response | 18 months
  Tthe proportion of patients who have a partial or complete response or stable disease(CBR) with Ribociclib at 18 months based on Response Evaluation Criteria in Solid Tumors RECIST v1.1
Ribociclib line of therapy treatment pattern | 18 months
  Ribociclib line of therapy treatment pattern at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, Muscat, Oman
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Al Ain Abu Dhabi, United Arab Emirates, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No